CLINICAL TRIAL: NCT03677531
Title: VidRT: Video Distraction During Radiation Therapy to Decrease Use of Pediatric Sedation
Brief Title: Video Distraction to Decrease Use of Sedation in Pediatric Participants During Radiation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jerry Jaboin, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00018053; NCI-2018-01505 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018053 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2018-09-14; First posted 2018-09-19 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy; Radiation; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Other (radiation therapy, videos) (Experimental): Participants undergo daily radiation therapy and watch videos/movies of their choice during treatments.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Other: Video

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Other: Video — Watch video of choice during RT

SUMMARY:
This phase I pilot trial studies how well video distraction works to decrease the use of sedation in pediatric participants during radiation therapy. Radiation treatment requires participants to lie very still (for accuracy). Many children cannot do this without sedation. Watching movies during radiation may distract children so they don't need sedation to complete treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the use of video distraction during radiation therapy (VidRT) during radiation for patients ages 3 to 13 decreases the rate of sedation use compared to patients previously treated without VidRT.

SECONDARY OBJECTIVE:

I. To determine which variables are associated with decreased need for sedation use. Variables will include patient age, length of treatment time (number of treatments and beam-on time), oncologic diagnosis, use of immobilization devices, pre-existing developmental or psychiatric diagnoses (attention deficit hyperactivity disorder [ADHD], dissociative disorders [DD], anxiety, depression, developmental delay, learning disability), pain scale ratings at time of first radiation treatment (0-10).

EXPLORATORY OBJECTIVES:

I. To determine the impact of VidRT on patient-reported quality of life prior to starting, during, and at the end of treatment using the pediatric quality of life inventory surveys including the Pediatric Quality of Life Inventory (PedsQL) - 4.0 Core and Peds QL- 3.0 brain tumor questionnaires.

II. To determine the impact of VidRT on patient-reported anxiety throughout radiation treatment as monitored by Patient-Reported Outcomes Measurement Information System (PROMIS) pediatric item bank version (v) 2.0 anxiety questionnaire.

III. To determine if workup assessment category for patient being low, medium, or high risk of needing sedation correlates to actual sedation use.

OUTLINE:

Participants undergo daily radiation therapy and watch videos/movies of their choice during treatments.

ELIGIBILITY:
Inclusion Criteria:

* All races and genders will be included.
* Patients with all tumor types will be included.

Exclusion Criteria:

* Patients < 3 years and > 13 years of age will be excluded.
* Patients with underlying movement disorders will be excluded.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Rate of sedation use calculated using number of treatment sessions | Up to 1 year
  A 1-sided binomial test will be used.

SECONDARY OUTCOMES:
Patient age and association with decreased sedation use | Up to 1 year
  A multivariate analysis will be used to determine which variables correlate with increased sedation use.
Number of treatments and association with decreased sedation use | Up to 1 year
  A multivariate analysis will be used to determine which variables correlate with increased sedation use.
Beam "on-time" and association with decreased sedation use | Up to 1 year
  A multivariate analysis will be used to determine which variables correlate with increased sedation use
Oncologic diagnosis and association with decreased sedation use | Up to 1 year
  A multivariate analysis will be used to determine which variables correlate with increased sedation use.
Use of immobilization device and association with decreased sedation use | Up to 1 year
  A multivariate analysis will be used to determine which variables correlate with increased sedation use.
Pre-existing developmental delay or psychiatric diagnosis and association with decreased sedation use | Up to 1 year
  A multivariate analysis will be used to determine which variables correlate with increased sedation use.
Pain at time of first radiation treatment and association with decreased sedation use (on a scale of one to ten) | Up to 1 year
  A multivariate analysis will be used to determine which variables correlate with increased sedation use.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry J Jaboin, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States